CLINICAL TRIAL: NCT04782440
Title: The Effect of Telerehabilitation of Patients With Duchenne Muscular Dystrophy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1455
Record Dates: First submitted 2021-03-02; First posted 2021-03-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation (Experimental)
  Interventions: Other: Telerehabilitaton
- Home exercise (Active Comparator)
  Interventions: Other: Home exercise

INTERVENTIONS:
Other: Telerehabilitaton — Patients will receive telerehabilitation sessions that include strengthening, stretching and range of motion exercises
  Arms: Telerehabilitation
Other: Home exercise — Patients will be given a home-based exercise program without telerehabilitation supervision
  Arms: Home exercise

SUMMARY:
The aim of this study is to investigate the effect of a telerehabilitation approach to patients with Duchenne Muscular Dystrophy and evaluate patients' motor function, parents' anxiety and depression levels before and after the intervention

ELIGIBILITY:
Inclusion Criteria:

* Patients with Duchenne muscular dystrophy

Exclusion Criteria:

* Patients without the ability of independent ambulation

Ages: 6 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Quick motor function test | 2 months

IPD SHARING:
Plan to Share IPD: Undecided